CLINICAL TRIAL: NCT02644837
Title: Randomised Crossover Comparison of the Ambu AuraGain and the iGel in Anaesthetised Adults
Brief Title: AuraGain and iGel Crossover Comparison
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful attempts to recruit participants
Sponsor: NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015AN07
Record Dates: First submitted 2015-12-04; First posted 2016-01-01 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Airway Management; Laryngeal Mask Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- i-Gel and AuraGain (Active Comparator): In this arm of the crossover study, patients will undergo insertion of Ambu AuraGain laryngeal mask airway and iGel and will undergo initial management with the iGel. Primary and Secondary outcomes will be assessed. The initial device will be removed and subsequent Airway management will then be undertaken with the Ambu AuraGain and the same outcomes will be assessed.
  Interventions with both devices will be
  1. Insertion of the laryngeal mask airway
  2. Assessment of ease of insertion
  3. Ability to perform positive pressure ventilation
  4. Measurement of OLP
  5. Fibreoptic assessment with Ambu A-scope
  6. Ability to insert nasogastric tube
  7. Record number of manipulations
  8. An assessment of device related trauma
  Interventions: Device: Insertion of Ambu AuraGain laryngeal mask airway and Igel; Device: Fibreoptic assessment with Ambu A-scope; Device: Ability to insert nasogastric tube; Device: Measurement of OLP; Device: Ability to perform positive pressure ventilation; Device: Assessment of ease of insertion; Device: Record number of manipulations; Device: Assessment of device related trauma
- AuraGain and i-Gel (Active Comparator): In this arm of the crossover study, patients will undergo insertion of the Ambu AuraGain laryngeal mask airway and i-Gel and will undergo initial management with the Ambu AuraGain.. Primary and Secondary outcomes will be assessed. Airway management will then be undertaken with the iGel device and the same outcomes will be assessed.
  Interventions with both devices will be
  1. Insertion of the laryngeal mask airway
  2. Assessment of ease of insertion
  3. Ability to perform positive pressure ventilation
  4. Measurement of OLP
  5. Fibreoptic assessment with Ambu A-scope
  6. Ability to insert nasogastric tube
  7. Record number of manipulations
  8. An assessment of device related trauma
  Interventions: Device: Insertion of Ambu AuraGain laryngeal mask airway and Igel; Device: Fibreoptic assessment with Ambu A-scope; Device: Ability to insert nasogastric tube; Device: Measurement of OLP; Device: Ability to perform positive pressure ventilation; Device: Assessment of ease of insertion; Device: Record number of manipulations; Device: Assessment of device related trauma

INTERVENTIONS:
Device: Insertion of Ambu AuraGain laryngeal mask airway and Igel — Insertion of Ambu AuraGain and iGel laryngeal mask airways in accordance with manufacturer instruction
Device: Fibreoptic assessment with Ambu A-scope — Passage of Ambu a-scope fibrescope down shaft of laryngeal mask airway and assessment of alignment with glottis in relation to amount of glottis that is easily visualised
Device: Ability to insert nasogastric tube — Passage of nasogastric tube down the gastric drainage channel of the device in accordance with manufacturer guidance
Device: Measurement of OLP — Measurement of OLP by closing the adjustable pressure limiting valve against a constant fresh gas flow rate of 3 litres/minute
Device: Ability to perform positive pressure ventilation — The ability to deliver 6 mls/kg volumes breaths by means of positive pressure ventilation will be assessed
Device: Assessment of ease of insertion — Ease of insertion will be subjectively assessed by operator in relation to presence and nature of resistance to insertion of the device
Device: Record number of manipulations — The number of manipulations/adjustments will be recorded for the second device only for the remainder of the device use during surgery until the patient wakes.
Device: Assessment of device related trauma — Observation and assessment of any trauma caused by the insertion of the first device used

SUMMARY:
This study will look at key performance indicators of 2 supraglottic airway devices in anaesthetised adults in a crossover manner.

DETAILED DESCRIPTION:
A supraglottic airway device (SAD), also referred to as laryngeal mask airway (LMA), is a medical device that maintains a patients airway, allowing unobstructed ventilation during anaesthesia. They are designed to sit in the patient's hypopharynx (throat), with their elliptical head forming a seal around the supraglottic structures (the patients "voice box"). They have been in common use since 1989, transforming anaesthetic practice and are now the predominant airway device within anaesthesia, being used in approximately 56% of all general anaesthetic cases in the UK(1). Their popularity for routine use stems from its perceived benefits over traditional forms of airway management coupled with their high overall success rate and low complication rate.

SADs, in anaesthetic practice, are inserted after induction of general anaesthesia, by or under supervision of, a trained medical professional. All patients are fully monitored as set out by the Association of Anaesthetist of Great Britain and Ireland; Recommendations for standards of monitoring during anaesthesia and recovery (2). Devices are used in concordance with manufacturer instruction. Successful first time placement is achieved in a large majority of patients and allows provision of oxygen and ventilation. In some patients, one device or size of device may present sub-optimal performance resulting in the removal of the device. Further actions in this scenario would include attempting a second insertion of the same device, attempting an insertion with an alternative size of the same device or a further attempt with an alterative design of device in order to achieve a patent airway. Further attempts may be taken but should be limited to avoid unnecessary trauma. In some cases the use of the SAD is abandoned and the patient is intubated with an endotracheal tube in order to provide a safe secure airway.

Alternatives to use of a SAD for airway management include use of a simple facemask or tracheal intubation with an endotracheal tube. Advantages of using a SAD for anaesthetic airway management compared to a facemask are improved oxygen saturation and less operator/anaesthetist fatigue. Compared to an endotracheal tube the advantages of using a SAD are improved haemodynamic stability at induction and emergence from anaesthesia, reduced anaesthetic requirements, improved quality of emergence, lower incidence of sore throat, increased ease of placement and reduced risk of dental damage. Risks of using an LMA compared to an endotracheal tube are increased gastric insufflation and aspiration with these being more common in patients who are poorly selected for anaesthesia with a SAD. Sore throat is the most common complication with a study

There have been significant developments in design in the SAD market in recent years with development of a "second generation" range of devices involving new materials and designs that integrate protective bite blocks, gastric drainage channels and improved supraglottic seal enhancing patient safety when using these devices. There are now some new "third generation" SADs on the market with designs that may enhance anaesthetic practice and improve patient safety further.

This study will follow similar ethically approved protocols used in published studies comparing airway equipment (3,4). These are only 2 examples but there are hundreds of LMA studies throughout the literature. The Ambu AuraGain is a new device and has not been studied fully. Comparative studies frequently assess oropharyngeal leak pressure (OLP), a fibre optic assessment of glottic alignment, ease of insertion, ability to insert a nasogastric tube down the gastric port and frequency of manipulations.

We propose a crossover design to better detect differences between the two devices as this eliminates confounding differences in patient characteristics and demographics.

There have been significant developments in design in the SAD market in recent years with

Our proposal would be to carry out a randomised crossover comparison between a new "third generation" SAD; the AuraGainTM (Ambu, Copenhagen, Denmark) and our current "second generation" SAD; the i-gel (Intersurgical Ltd, Wokingham, UK) to examine and compare key performance indicators with their use.

The AuraGain is a new device on the market and has not been compared to other devices yet.

ELIGIBILITY:
Inclusion Criteria:

* patients who have read and understood patient information leaflets about the study and undergo informed consent.
* patients whose anaesthesia management is being carried out by one of the named investigators
* adult (age >18 years) patients undergoing general anaesthesia
* American Society of Anaesthesiology Grading (ASA) 1-3
* suitability for general anaesthesia using a laryngeal mask airway device

Exclusion Criteria;

* the presence of significant acute or chronic lung disease
* pathology of neck or upper respiratory tract
* an identified or anticipated difficult intubation
* an increased risk of aspiration (hiatus hernia, gastro-oesophageal reflux or full stomach etc.) pregnant women
* a body mass index greater than 35kg.m-2
* patients unable to communicate fully in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | Up to 3 minutes of successful insertion of each device
  If successful ventilation is achieved with the device, the investigator will measure OLP by closing the Adjustable Pressure Limiting valve on the anaesthetic machine; with a fresh gas flow of 3l/min. Pressure at which equilibrium is reached will be deemed the OLP. Pressure will not be allowed to exceed 40cmH20.

SECONDARY OUTCOMES:
Ease of insertion | Up to 1 minute on each insertion attempt
  Subjective assessment of ease of insertion of device
Number of attempts required to insert | Up to 1 minute of completion of total insertion attempts
  Record of number of attempts required to insert successfully
Evidence of Airway Trauma | Up to 1 minute after removal of first device used
  Examination of device for signs of airway trauma produced during insertion of first device
Adequacy of positive pressure ventilation | Up to 1 minute after successful insertion of device and after completion of outcome 4 measurement
  • Adequacy of ventilation as assessed by the presence of square wave capnography indicative of unobstructed ventilation and the ability to provide chest wall movement that approximates to the patients normal tidal volume
Fibreoptic assessment of device position | Up to 5 minutes after successful insertion and after completion of outcome 5 measurement
  A fibreoptic scope will be inserted down the shaft of each device, whilst ventilation continues and a subjective assessment of alignment with glottic structures is made.
Ability to insert nasogastric tube down gastric channel of device | Up to 5 minutes after successful insertion and after completion of outcome 6 measurement
Intraoperative manipulations required | For up to 2 hours after induction of anaesthesia
  Intraoperative manipulations during procedure recorded for second device only

CONTACTS AND LOCATIONS:
Overall Officials: Simon M Crawley, MBChB FRCA, Principal Investigator — Consultant Anaesthetist
Locations (1):
- Ninewells Hospital, Dundee, Angus, United Kingdom

IPD SHARING:
Plan to Share IPD: No